CLINICAL TRIAL: NCT04779996
Title: Antibodies Production After Covid-19 Vaccination Among Patients With Medical History of Cancer and Anti-CD-20 Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Auxilio Mutuo Cancer Center (Other)
Responsible Party: Principal Investigator, Fernando Cabanillas, Fernando Cabanillas, MD, Auxilio Mutuo Cancer Center
Other Study IDs: CCAM 21-01
Record Dates: First submitted 2021-03-02; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Cancer; HIV Infections
MeSH Terms: conditions — COVID-19; Neoplasms; HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Laboratory Samples — 1. After full vaccination with a Covid 19 vaccine, the following laboratory samples will be taken one time only, two weeks after full dose vaccination: i. Serologic rapid test (IgG, IgM) ii. Serum quantitative immunoglobulin levels iii. CD4 level iv. CD8 level
  2. Laboratory samples will be taken at Hospital Auxilio Mutuo Laboratorio Clínico. Likewise, the Immuno Reference Lab might be used as an alternative.
  3. Since monoclonal antibody therapy can induce hypogammaglobulinemia, we will measure gammaglobulin levels to correlate with antibody response to vaccine. Similarly, we will evaluate the CD4 and CD8 counts.

SUMMARY:
This is a Phase II study designed to investigate if the Covid 19 vaccines are capable of eliciting production of antibodies against S protein of Sar-S-Cov-2 virus among patients with medical history of cancer previously treated with monoclonal anti CD-20 antibodies. The antibody production is defined based on the detection of antibodies in the serologic Covid-19 rapid test against S protein or with semiquantitative assay when it becomes available.

ELIGIBILITY:
Inclusion Criteria:

* All patients either diagnosed with cancer or with HIV positivity or treated with an antineoplastic regimen including anti CD-20 after Covid-19 vaccine will be registered on the study regardless of their type of cancer or type of antineoplastic regimen.
* Patients 21 years or older diagnosed with cancer treated with antineoplastic regimen or anti CD-20, or with HIV infection vaccinated with 2 doses of anti Covid-19 vaccine.
* Eligible patients will be registered on study after a Covid -19 vaccine has been scheduled.
* In order to be screened for Covid 19 antibodies, they must be tested at least two weeks after the second dose of Covid-19 vaccination.

Exclusion Criteria:

* Anyone who has not been treated with anti-CD20 antibodies or with chemotherapy who doesn't have HIV infection or who has not received chemotherapy for cancer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients either diagnosed with cancer or with HIV positivity or treated with an antineoplastic regimen including anti CD-20 after Covid-19 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Two weeks after full dose vaccination.
  To determine if patients with cancer history or HIV positivity previously treated with monoclonal anti CD-20 are able to produce antibodies after Covid-19 vaccination.
  a. Antibody Production defined as: 1. Positive serologic Covid-19 antibodies rapid test against S protein.

SECONDARY OUTCOMES:
Secondary objective 1 | Two weeks after full dose vaccination.
  Evaluate the Correlation of immunoglobulin levels and the development of Covid-19 antibodies.
Secondary objective 2 | Two weeks after full dose vaccination.
  Evaluate the correlation of CD4/CD8 counts with the development of Covid-19 antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker D, Roberts CAK, Pryce G, Kang AS, Marta M, Reyes S, Schmierer K, Giovannoni G, Amor S. COVID-19 vaccine-readiness for anti-CD20-depleting therapy in autoimmune diseases. Clin Exp Immunol. 2020 Nov;202(2):149-161. doi: 10.1111/cei.13495. Epub 2020 Aug 1. PMID 32671831
- [Background] Houot R, Levy R, Cartron G, Armand P. Could anti-CD20 therapy jeopardise the efficacy of a SARS-CoV-2 vaccine? Eur J Cancer. 2020 Sep;136:4-6. doi: 10.1016/j.ejca.2020.06.017. Epub 2020 Jun 25. PMID 32619884
- [Background] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735
- See also: OpenSAFELY: factors associated with COVID-19-related hospital death in the linked electronic health records of 17 million adult NHS patients. — https://www.medrxiv.org/content/10.1101/2020.05.06.20092999v1